CLINICAL TRIAL: NCT01141699
Title: A Study of Compliant Behaviors and Associated Factors of Women Breast Screening in the Shuang Ho Region of Taipei City.
Brief Title: A Study of Compliant Behaviors and Associated Factors of Women Breast Screening
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Head Nurse of Cancer Center, Cancer Center of Taipei Medical University WanFang Hospital
Other Study IDs: IRB99006
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Health Behaviors
Keywords: women health behaviors
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- female: Women who live in the Shuang Ho Region of Taipei City. Women can read and write chinese language.

SUMMARY:
There were a breast cancer screening activity in Taipei Medical University-Shuang Ho Hospital. We did an intervention with woman who joined the activity.The most important part in the intervention was to know health behavior about the breast cancer prevention.By doing the study, the investigators will know how to promote the health activity in our community.

DETAILED DESCRIPTION:
When the investigators get these women's health behavior imagination, the investigators can know how much breast cancer screening activity do these people have. The most important part for us is to understand how to promote health behavior to women who live around Shuang area.

ELIGIBILITY:
Inclusion Criteria:

1. women
2. can read words

Exclusion Criteria:

NA

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The women live in the Shuang Ho Region of Taipei City
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shing-Fang Wang, Principal Investigator — Cancer Center of Taipei Medical University Shuang Ho Hospital